CLINICAL TRIAL: NCT02788357
Title: Enhancement of Post-stroke Neural Plasticity With Atomoxetine: a Pilot Study
Brief Title: Post-stroke Neural Plasticity With Atomoxetine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumy Sawaki (Other)
Responsible Party: Sponsor-Investigator, Lumy Sawaki, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: No ID
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Atomoxetine Hydrochloride; Placebos
Keywords: motor training; motor recovery; human; neuroplasticity; transcranial magnetic stimulation
MeSH Terms: interventions — Atomoxetine Hydrochloride; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine with motor training (Experimental): 40 mg atomoxetine paired with task-oriented therapy for 10 consecutive weekdays
  Interventions: Drug: Atomoxetine
- Placebo with motor training (Placebo Comparator): Placebo capsules paired with task-oriented therapy for 10 consecutive weekdays
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Subjects will receive a single daily oral dose of 40 mg of atomoxetine. We will administer 2 hours/daily of motor training sixty minutes after drug intake.
  Other Names: Strattera
  Arms: Atomoxetine with motor training
Drug: Placebo — Subjects will receive a single daily oral dose of placebo. We will administer 2 hours/daily of motor training sixty minutes after drug intake.
  Other Names: Sham
  Arms: Placebo with motor training

SUMMARY:
This proposal evaluates the safety and effectiveness of a noradrenergic drug named atomoxetine combined with motor training to enhance cortical plasticity and improve hand function after stroke.

DETAILED DESCRIPTION:
Extensive studies in laboratory animals and humans over the last ten years indicate that some medications, especially amphetamine, given with specific physical therapy may improve motor learning (and therefore recovery from stroke) more than physical therapy alone. However, the number of patients in clinical trials who have received physical therapy and amphetamine is very small, for two reasons: because amphetamine may interact with many other medications that stroke patients are already taking, and because its potential for addiction precludes its use on a daily basis. The investigators now wish to evaluate the effectiveness of a more selective medication, atomoxetine, known to have many fewer side effects and no potential for drug addiction. The proposed mechanism by which amphetamine enhances recovery is by increasing central levels of norepinephrine. While the investigators already know that this drug is more selective than amphetamine, the investigators would like to evaluate its effects on hand motor learning and motor recovery in chronic stroke patients in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients
* Single stroke
* Chronic (more than 6 months after from stroke)
* At least 21 years old, but there is no upper age range for this project.
* Participants NOT able to extend the affected metacarpophalangeal joints at least 10° and the wrist 20°.

Exclusion Criteria:

* History of head injury with loss of consciousness
* History of severe alcohol or drug abuse
* History of psychiatric illness
* Unstable cardiac dysrhythmia
* High blood pressure (systolic pressure >160 mm Hg and/or diastolic pressure >100 mm Hg)
* History of myocardial infarction or unstable angina
* Pregnancy
* Glaucoma, history of hypersensitivity or idiosyncrasy to sympathomimetic drugs.
* Subjects using drugs suspected of interfering with plasticity, such as MAOI, alpha-adrenergic antagonists, benzodiazepines, muscarinic receptor antagonists, dopaminergic antagonists, or other neuroleptics within 3 months of recruitment.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ward A, Carrico C, Powell E, Westgate PM, Nichols L, Fleischer A, Sawaki L. Safety and improvement of movement function after stroke with atomoxetine: A pilot randomized trial. Restor Neurol Neurosci. 2017;35(1):1-10. doi: 10.3233/RNN-160673. PMID 27858723

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atomoxetine With Motor Training | Placebo With Motor Training
Started | 6 | 6
Completed | 3 | 6
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine With Motor Training | Placebo With Motor Training | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (12.6) | 59.8 (5.2) | 55.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Fugl Meyer Assessment
Description: Score after intervention minus baseline score, score at 1-month follow-up minus baseline score. The possible scores range from 0 to 66, with 66 indicating the best performance.
Time Frame: baseline, post-intervention, 1-month follow-up
Population: 3 subjects in Atomoxetine group were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine With Motor Training | Placebo With Motor Training
Number analyzed (Participants) | 6 | 6
units on a scale
  Post-intervention minus baseline | 9.3 [5.4 to 13.2] | 2.2 [-1.7 to 6.1]
  1-month follow-up minus baseline: number analyzed (Participants) | 3 | 6
  1-month follow-up minus baseline | 11.9 [5.9 to 17.9] | 5.8 [1.5 to 10.2]

2. Secondary Outcome: Change in Action Arm Research Test (ARAT)
Description: Score at post-intervention minus baseline, score at 1-month follow-up minus baseline. The score is calculated by summing the scores for 19 individual tasks. The possible scores range from 0 to 57, with higher scores indicating better performance.
Time Frame: baseline, post-intervention, 1-month follow-up
Population: 3 subjects in the Atomoxetine group were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine With Motor Training | Placebo With Motor Training
Number analyzed (Participants) | 6 | 6
units on a scale
  Post-intervention minus baseline | 7.7 [4.6 to 10.7] | 5.3 [2.3 to 8.4]
  1-month follow-up minus baseline: number analyzed (Participants) | 3 | 6
  1-month follow-up minus baseline | 10.1 [5.1 to 15.1] | 6.5 [2.6 to 10.4]

3. Secondary Outcome: Change in Wolf Motor Function Test (WMFT)
Description: Score at post-intervention minus baseline, score at 1-month follow-up minus baseline. Each task is scored as amount of time taken to complete a task, which may range from just over 0 to 120 seconds. If the subject is unable to complete the task within 120 seconds, a score of 121 seconds is given. The scores from the 15 individual tasks are averaged, then the log is taken, resulting in the overall score. Therefore, the larger the score, the longer required to perform the tasks. Negative changes in score indicate that a subject, on average, was able to complete the tasks faster at post-intervention or at 1-month follow-up than at baseline.
Time Frame: baseline, post-intervention, 1-month follow-up
Population: 3 subjects in the Atomoxetine group were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: log(seconds)
Arm/Group | Atomoxetine With Motor Training | Placebo With Motor Training
Number analyzed (Participants) | 6 | 6
log(seconds)
  Post-intervention minus baseline | -0.1 [-0.26 to 0.06] | -0.19 [-0.35 to -0.03]
  1-month follow-up minus baseline: number analyzed (Participants) | 3 | 6
  1-month follow-up minus baseline | -0.11 [-0.28 to 0.06] | -0.2 [-0.37 to -0.04]

4. Secondary Outcome: Transcranial Magnetic Stimulation
Time Frame: Score change after 10 days of intervention compared to baseline; Score change after 1-month after the intervention compared to baseline
Population: This data is not available at this time, as a relocation occurred during the project. Data collected at the previous institution used different software and stored the data in a different format than is currently used. Therefore, reconciliation of this data is being attempted at this time.
Arm/Group | Atomoxetine With Motor Training | Placebo With Motor Training
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Atomoxetine With Motor Training | Placebo With Motor Training
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No